CLINICAL TRIAL: NCT05439252
Title: The Acceptability of Exercise Snacking to Improve Leg Strength in Memory Clinic Outpatients: a Pilot Study
Brief Title: Exercise Snacking to Improve Strength and STability: ESISST Pilot Study
Acronym: ESSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Dr Oliver Perkin, Principle Investigator, University of Bath
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UoB-ESS-02
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Acceptability of an Exercise Intervention
Keywords: Exercise Snacking; Elderly; Homebased exercise; Outpatient

STUDY DESIGN:
Intervention Model Description: Single group, pre-test-post-test pilot study of acceptability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Snacking Group (Experimental): For 28 days, this group will be asked to perform two 'exercise snacks' a day; once in the morning and once in the evening, and record exercise snacking compliance data in a log book
  Interventions: Behavioral: Exercise Snacking

INTERVENTIONS:
Behavioral: Exercise Snacking — Each bout of exercise snacking consists of 5 exercise. Each exercise is performed for one minute, with aim of completing as many repetitions as possible of that exercise in that minute. One minute of rest is observed between each exercise of the exercise snack. The five exercises are sit-to-stand from a chair, seated overhead arm raises, march on the spot, seated arm raises and shoulder touches, and seated calf raises. The sit-to-stand exercise is always performed first, with the number of repetitions achieved recorded, and subsequent exercises performed in any order without recording of repetitions.

SUMMARY:
As we age, muscles can become progressively weaker to the point that tasks of daily living cannot be carried out safely. However, regular resistance exercise training has been shown to maintain and even increase muscle strength in older adults. Previous research has identified a homebased, non-loaded, lower limb only, 'exercise snacking' model that does not require exercise equipment or supervision as a viable alternative exercise strategy to traditional resistance exercise, with potential to improve leg muscle strength in healthy older adults. This approach has been shown to be feasible and acceptable to general healthy older adult population, however this approach to exercise focussed on improving strength has not been considered in a clinical population.

This research seeks to investigate the acceptability of 28 days of homebased exercise snacking in outpatients with attending the memory clinic at the Research Institute for Care of the Elderly (RICE) Centre in Bath, UK, with diagnosis limited to mild cognitive impairment only. This study will improve understanding of how zero-cost exercise strategies to potentially improve muscle function and delay frailty could be incorporated in daily routines of older adults.

DETAILED DESCRIPTION:
Potential participants will be identified by clinicians during memory clinic outpatient appointments at the Research Institute for Care of the Elderly (RICE) in Bath. Clinicians will provide a brief overview of the study, and the Participant Information sheet to those individuals interested in participating.

Potential participants will then be contacted by the researcher at RICE to arrange a screening meeting. This will be a face-to-face meeting, taking place at RICE. Potential participants are invited to bring carers to this meeting.

At the screening meeting, a verbal overview of the study will be provided by the researcher and written informed consent must be provided by the potential participant after they have had chance to ask questions about the study.

A health screen questionnaire will be completed, and basic cognitive and physical function tests will be undertaken to assess participant eligibility. Participants passing these tests will be invited to participate.

Eligible participants will be asked to complete questionnaires and undertake further tests of physical function, including a thorough practice of the exercise intervention. The baseline assessment will take place during the same visit as the screening meeting. If the researcher believes that performance in these baseline physical function tests indicates that it would not be safe for the participant to continue in the study, then then will be withdrawn at that point.

All participants will be asked to undertake 28 consecutive days of exercise snacking. This involves two bouts of exercise per day, one in the morning and one in the afternoon/evening. Each bout will consist of five exercises, with each exercise performed for 60 seconds only, followed by 60 seconds of rest, before performing the next exercise. The exercises require no specialist equipment or clothing but must only be performed when there is someone else in the house that would be capable of calling for help in the event of an emergency.

Participants will be provided with a logbook to record information about each exercise bout, and an appendix document with detailed instruction on how to perform exercise snacking. Participants will also be asked to wear a physical activity monitor for the first seven days of exercise snacking, and to return this in a pre-paid and addressed envelope after this period of wear.

Participants will be invited to the RICE centre within five days completing the exercise snacking intervention to complete the same questionnaires and physical function tests that were undertaken at the baseline assessment. A further questionnaire exploring the acceptability of the exercise snacking intervention will be completed. Participants will also be invited to undertake a qualitative interview with the researcher to gain further insight into the participant's experience of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged >65 years
* Have attended the Memory Clinic at the RICE Centre in Bath
* Mini-mental state examination (MMSE) score of ≥20
* Short Physical Performance Battery (SPPB) score 3-8 and not scoring 0 on any component of the test
* Capability to safely perform the exercise snacking movements, assessed by a researcher during screening, and be able to have someone present in the home who could call for help if required during all exercise snacks.
* Not regularly engaging in recreational sports or structured exercise (once a week or more).
* Have a foreseeable clear period of 28 consecutive days in which to perform the exercise snacking protocol (i.e. no planned holidays or hospitalisation)

Exclusion Criteria:

* Co-morbidity preventing participation (e.g. severe breathlessness, pain, psychosis, Parkinson's, Dementia with Lewy Bodies, or other severe neurological disease)
* Individuals with a history of bone, joint or neuromuscular problems or a current musculoskeletal injury ascertained through preliminary screening that would prevent exercise snacking or be made worse by performing exercise snacking.
* Individuals with contraindications to exercise including chest pain, dizziness, or loss of consciousness, or who have been instructed by their doctor to only do physical activity recommended by them.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Welsh, MD, PhD, Study Director — RICE
Locations (1):
- University of Bath, Bath, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Western MJ, Welsh T, Keen K, Bishop V, Perkin OJ. Exercise snacking to improve physical function in pre-frail older adult memory clinic patients: a 28-day pilot study. BMC Geriatr. 2023 Aug 4;23(1):471. doi: 10.1186/s12877-023-04169-6. PMID 37542234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This pilot study aimed to collect primary outcome measure from 20 participants in a single group study design. Participants were all outpatients who had attended an NHS commissioned memory clinic in Bath, UK. All data collection took place during a three-month testing window, with a rolling recruitment strategy capped at up to 10 replacement participants who could complete the 28-day intervention and associated assessments within the three-month testing phase.
Pre-assignment Details: The baseline assessment took place during the same visit as the screening, provided that potential participants met all eligibility criteria and enrolled in the study, and there was no group assignment as this was a single group study design.
Period: Overall Study
Arm/Group | Exercise Snacking Group
Started | 21
Completed | 18
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Outpatients aged >65 years who had attended an NHS commissioned memory clinic at the Research Institute for Care of Older Adults in Bath, UK
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 20
  Asian British | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 21

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Intervention
Description: Participants will be asked to complete a Theoretical Framework of Acceptability questionnaire on their experiences of the exercise snacking questionnaire.
  The scale scores range from 0 to 5 with high scores indicating greater acceptability, and the total score representing the mean average of 7 individual domains of acceptability (each also rated 0-5).
Time Frame: 28-days (post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale | 4.6 (0.6)

2. Secondary Outcome: Attitudes to Exercise
Description: Outcome Expectancy for Exercise Questionnaire Score on a scale of 0-5, with higher scores indicating higher outcome expectancy
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 4.0 (0.6)
  Post-intervention | 4.3 (0.5)

3. Secondary Outcome: Self-confidence for Exercise
Description: The 'Barriers Self-Efficacy Scale', (BARSE), to assess participants perceived capabilities to exercise. The scale ranges from 0-100, with a higher score indicating higher self-efficacy.
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 70.1 (26.2)
  Post-intervention | 66.3 (16.3)

4. Secondary Outcome: Psychological Need Satisfaction for Exercise
Description: Psychological need satisfaction for exercise questionnaire Score on a scale of 0-6, with higher scores indicating a greater satisfaction of basic psychological needs
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 5 (0.7)
  Post-intervention | 5 (.7)

5. Secondary Outcome: Current Mental Health
Description: Patient Health Questionnaire Score on a scale of 0-27, with lower scores indicating less depression
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 3.5 (3.5)
  Post-intervention | 3.7 (3.7)

6. Secondary Outcome: Patient Anxiety
Description: Generalised Anxiety Disorder Assessment Score on a scale of 0-21, with lower scores indicating lower anxiety
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 2 (2)
  Poat-intervention | 1.6 (2.1)

7. Secondary Outcome: General Health
Description: Short Form Health Survey (SF-36) Separate scales from 0 to 100 for each of the two domains (physical and mental), with higher scores meaning better health status in both. The two domains are reported separately but not combined.
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Physical Domain: Baseline | 48.5 (8.0)
  Physical Domain: Post-Intervention | 46.1 (6.8)
  Mental Domain: Baseline | 47.5 (11.9)
  Mental Domain: Post-intervention | 51.3 (12.8)

8. Secondary Outcome: Patient Vitality
Description: Subjective Vitality Index Score on a scale of 0-49, with higher scores indicating greater vitality
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 30.8 (8.7)
  Post-intervention | 32.4 (6.1)

9. Secondary Outcome: Patient Life Satisfaction
Description: Life Satisfaction Scale Score on a scale of 0-35, with higher scores indicating greater satisfaction with life
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 29 (4.1)
  Post-intervention | 27.7 (5.5)

10. Secondary Outcome: Patient Quality of Life
Description: Overall quality of life scale Score on a scale of 0-100, with higher scores indicating better quality of life
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 82.5 (11.1)
  Post-intervention | 79.4 (8.2)

11. Secondary Outcome: Cognitive Assessment
Description: Montreal Cognitive Assessment Score on a scale of 0-30, with lower scores indicating greater cognitive impairment
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 23.3 (4.0)
  Post-intervention | 24.3 (4.0)

12. Secondary Outcome: Cognitive Assessment
Description: Groningen Frailty Index Score on a scale of 0-15, with higher scores being more frail
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 3.9 (2.1)
  Post-intervention | 3.6 (1.9)

13. Secondary Outcome: Physical Function Assessments
Description: Short Physical Performance Battery Score on a scale of 0-12, with higher scores indicating greater physical function
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 7 (1.5)
  Post-intervention | 8.8 (2.3)

14. Secondary Outcome: Physical Function Assessments
Description: 60 second sit-to-stand test The number of sit-to-stands completed in 60 seconds
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: repetitions completed
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
repetitions completed
  Baseline | 17.2 (4.9)
  Post-intervention | 22.7 (7.4)

15. Secondary Outcome: Physical Function Assessments
Description: 60 second sit-to-stand rating of perceived exertion Borg scale from 6-20, with higher scores indicating greater perceived exertion
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 10.8 (2.1)
  Post-intervention | 11.6 (2.0)

16. Secondary Outcome: Physical Function Assessments
Description: Standing balance test scores Maximum time for single leg balance holds, capped at 60 seconds on each leg
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
seconds
  Right leg; Baseline | 27.3 (24.5)
  Right leg; Post-intervention | 26.9 (21.9)
  Left leg; Baseline | 22.1 (21.2)
  Left leg; Post-intervention | 28.8 (22.4)

17. Secondary Outcome: Physical Function Assessments
Description: Timed-up-and-go Time in seconds to complete a functional movement task
Time Frame: 28-days (pre-to-post intervention)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Exercise Snacking Group
Number analyzed (Participants) | 18
time in seconds
  Baseline | 12.6 (5.0)
  Post-intervention | 10.8 (5.1)

18. Other Pre Specified Outcome: Acceptability of the Intervention
Description: OPTIONAL qualitative exit interview
Time Frame: 28-days (post intervention)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning of screening to the end of the final assessment, with final assessment scheduled within two weeks of completing the 28-day intervention which began at the screening session. Thus the time period for adverse event collect was 4-6 weeks.
Description: Adverse events were as per the definitions from clinicaltrials.gov
Arm/Group | Exercise Snacking Group
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT05439252/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT05439252/ICF_001.pdf